CLINICAL TRIAL: NCT05386901
Title: The Effects of Individualized Lung-protective Ventilation With Lung Dynamic Compliance-guided Positive End-expiratory Pressure(PEEP) Titration on Postoperative Pulmonary Complications of Pediatric Video-assisted Thoracoscopic Surgery
Acronym: PEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiaxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Jiaxiang Chen, Postgraduate Student, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13229547507
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Surgery
Keywords: Lung dynamic compliance; Positive end-expiratory pressure(PEEP); One-lung ventilation(OLV); Lung protection strategy; Postoperative pulmonary complications(PPCs)

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to lung dynamic compliance-guided individualized PEEP group and traditional PEEP group.The traditional lung protective ventilation experimental group kept PEEP at 5cmH2O, and the lung dynamic compliance-oriented individualized PEEP group passed the incremental PEEP (0-14cmH2O). lung dynamic compliance==Vt/(Pplat-PEEP).The initial PEEP is set to 0cmH2O, and the PEEP is increased by 2cmH2O every 2 minutes. Observe the PEEP value corresponding to the maximum lung dynamic compliance during the process. After the incremental PEEP process is completed, set the PEEP value for ventilation until the end of the operation.
Who Masked: Participant
Masking Description: This experiment adopts a single-blind scheme. Only the researcher understands the grouping situation, and the research subjects do not know whether they are the experimental group or the control group. The researcher can better observe and understand the research subjects, and can timely and appropriately deal with possible occurrences of the research subjects when necessary. Unexpected problems, so that the safety of the research object is guaranteed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional positive end-expiratory pressure(PEEP) (Experimental): Once the patient is intubated and after initiating ventilation in a pressure control mode(PCV) using an airway pressure of 20-25mmHg with tidal volume not exceeding 6ml/kg of predicted body weight (PBW) and an inspiration: expiration ratio of 1:2;a respiratory rate of 20-30 breaths per minute to maintain the etCO2 at 35-40 mmHg.The investigators will set the PEEP value to 5 cmH2O until the end of the operation.
  Interventions: Procedure: Conventional positive end-expiratory pressure(PEEP)
- Lung dynamic compliance guided positive end-expiratory pressure(PEEP) (Experimental): Once the patient is intubated and after initiating ventilation in a pressure control mode(PCV) using an airway pressure of 20-25mmHg with tidal volume not exceeding 6ml/kg of predicted body weight (PBW) and an inspiration: expiration ratio of 1:2;a respiratory rate of 20-30 breaths per minute to maintain the etCO2 at 35-40 mmHg.The investigators will set initial PEEP to 0cmH2O,and the PEEP is increased by 2 cmH2O every 2 minutes.Observing the PEEP value corresponding to the maximum lung dynamic compliance during the process that lung dynamic compliance=Vt/(Pplat-PEEP).After the incremental PEEP process is completed, setting the PEEP value for ventilation until the end of the operation.
  Interventions: Procedure: Lung dynamic compliance guided positive end-expiratory pressure(PEEP)

INTERVENTIONS:
Procedure: Conventional positive end-expiratory pressure(PEEP) — Positive end-expiratory pressure is the mechanical ventilator that generates positive pressure during the inspiratory phase to pass gas into the lungs. When the airway opens at the end of expiration, the airway pressure remains above atmospheric pressure to prevent the alveoli from shrinking and collapsing.In this intervention arm It will be set to 5 cmH2O until the end of the operation.
  Arms: Conventional positive end-expiratory pressure(PEEP)
Procedure: Lung dynamic compliance guided positive end-expiratory pressure(PEEP) — Positive end-expiratory pressure is the mechanical ventilator that generates positive pressure during the inspiratory phase to pass gas into the lungs. When the airway opens at the end of expiration, the airway pressure remains above atmospheric pressure to prevent the alveoli from shrinking and collapsing.In this intervention arm It will be set to individual value until the end of the operation.The individualized values are obtained by observing the maximum Lung dynamic compliance during PEEP titration.
  Arms: Lung dynamic compliance guided positive end-expiratory pressure(PEEP)

SUMMARY:
This study evaluates the influence of individualized lung-protective ventilation strategy(LPVS) on postoperative pulmonary complications(PPCs) through a randomized controlled trial when children undergoing thoracoscopic surgery with one-lung ventilation(OLV).The investigators evaluate the impact of using lung dynamic compliance-guided Positive End-expiratory Pressure(PEEP) versus conventional PEEP on a pressure-controlled ventilation(PCV).The researchers also analyzed perioperative vital signs and respiratory indicators of these LPVS.

DETAILED DESCRIPTION:
With the advancement of pediatric thoracic surgery techniques, the age group of children who can receive thoracoscopic surgery is getting younger and younger, and even neonates can accept it. In thoracic surgery, the incidence of PPCs is as high as 30%-50%, which is one of the main reasons for poor prognosis, increased mortality and prolonged hospitalization. In recent years, more and more studies have shown that the perioperative implementation of appropriate LPVS can reduce the occurrence of PPCs. How to optimize the lung protection strategy in pediatric thoracic surgery has become one of the key issues of perioperative medical attention, and there is no consensus in clinical application.

LPVS is one of the important components of lung protection strategies, including low tidal volume, PEEP and lung recruitment strategies.How to choose the most suitable PEEP is an important part in the implementation of LPVS. The optimal PEEP value should be the corresponding pressure value when the compliance between alveolar opening and over-inflation is the best. In recent years, many scholars have studied PEEP titration methods, such as lung dynamic compliance-guided PEEP, pressure-volume (P-V) curve-guided PEEP, transpulmonary pressure-guided PEEP, and electrical impedance tomography (EIT)-guided PEEP and so on.However, there are no published studies addressing the effects of lung dynamic compliance-guided PEEP on PPCs and perioperative vital signs and respiratory indicators of pediatric surgical patients when associated with OLA strategies for ventilation.

This study is a randomized controlled trial. After meeting the inclusion conditions, the researchers were assigned to any of the two groups of lung dynamic compliance-guided individualized PEEP and conventional PEEP. The clinical anesthesia and mechanical ventilation parameter settings and data statistical analysis were completed by different anesthesiologists and participants.

On the day of surgery, standard monitoring was initiated on arrival in the theatre, including electrocardiography, pulse oximetry, and noninvasive blood pressure monitoring.Both groups were given routine standard anesthesia induction: intravenous injection of midazolam at 0.05-0.1 mg/kg of predicted body weight (PBW), propofol at 2-4 mg/kg of PBW, and intravenous injection of Sufentanil at 0.3-0.5 ug/kg of PBW, rocuronium at 0.5-1mg/kg of PBW.After adequate pre-oxygenation, endotracheal intubation and bronchial occluder placement under video laryngoscope, using fiberoptic bronchoscopy and auscultation make sure the occluder is properly positioned. The investigators will adjust breathing parameters after starting double-lung ventilation,which is a pressure control mode(PCV) using an airway pressure of 20-25mmHg with tidal volume not exceeding 6ml/kg of PBW and an inspiration: expiration ratio of 1:2;a respiratory rate of 20-40 breaths per minute to keep PaCO2 < 60 mmHg as well as FiO2 of 50% and flow of 3L/min.Then, the first lung recruitment strategy was started. The manual lung recruitment method was used, and the ventilation mode was manually controlled. The APL valve was adjusted to 30cmH2O, maintained for 15-20 seconds, and then returned to the machine-controlled ventilation mode. Arterial puncture and catheterization were performed to establish an invasive arterial monitoring channel. Intraoperative maintenance medication: 2%-3% sevoflurane, dexmedetomidine (0.1-0.2ug/kg.h of PBW), sufentanil and rocuronium bromide were added in stages according to intraoperative conditions to maintain sufficient doses above sedative analgesia and muscle relaxation.

Before starting OLV, pure oxygen hyperventilation was used, FiO2 was adjusted to 100%, and the maintenance time was not less than 3 minutes to increase the oxygen concentration in both lungs and improve the tolerance of children to hypoxia and the success rate of lung collapse. After switching to OLV, a second manual recruitment strategy was performed. The PEEP settings were divided into two groups: the canventional lung protective ventilation experimental group held PEEP at 5 cmH2O, the pulmonary dynamic compliance guided PEEP group passed increasing PEEP (0-14 cmH2O), and the lung dynamic compliance = Vt/(Pplat-PEEP).The initial PEEP is set to 0cmH2O, which is increased by 2 cmH2O every 2 minutes. Observe the PEEP value corresponding to the maximum lung dynamic compliance during the process. After the incremental PEEP process is completed, setting the PEEP value for ventilation until the end of the operation.

At the end of one-lung ventilation, a third manual recruitment maneuver was performed before switching to double-lung ventilation. After the operation, the patients were sent to the ICU with a tracheal catheters or sent to the PACU before extubation according to the condition of the child.

All data were collected, aggregated and maintained by a single investigator. Including preoperative demographic data, ARISCAT score data, surgery-related data, anesthesia-related data, intraoperative general vital signs and respiratory indicators, postoperative PPCs-related data, postoperative medication, other postoperative complications, hospital stay, ICU Hospitalization time, respiratory support time, hospitalization time, biochemical indicators during hospitalization, inflammatory indicators, electrolytes, cardiac function indicators, etc.

This study was a superiority test, so a one-sided test was used, and the first-class error (α) was set to 0.05, and the second-class error (β) was set to 0.2 (that is, the power of 1-β was set to 0.8). The main observation index of this study is the incidence of PPCs. According to the literature review, the incidence of PPCs in the two groups in similar studies was 11% and 39%, respectively. In PASS 15.0, "Test for Two Proportions" was selected for calculation. The dropout rate is set to 10%, and the calculation result is that each group needs 30 patients.It would be necessary to recruit 60 patients in the study.

The full analysis set was used for analysis. According to the basic principle of Intention-to-Treat (ITT), the analysis of the main indicators includes all randomized subjects, regardless of whether they completed the trial or not, that is, subjects who were lost to follow-up should also be included in the statistical analysis. Statistical software SPSS 26.0 was used for data processing and statistical analysis. Shapiro-Wilk test was first performed on the data, and continuous variable data (such as blood pressure, heart rate, driving pressure, oxygenation index, etc.) were determined to use t test or Mann-Whitney U test according to their normal distribution. Categorical variables (such as age, incidence of PPCs, etc.) were tested by χ² test, Fisher's exact test, and the results were expressed as mean ± standard deviation (SD), percentage (%) or median (interquartile range, IQR), P <0.05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing elective thoracoscopic pulmonary surgery.
* Written informed consent.
* Children under 5 years old (including 5 years old)
* ASA classification 1-2
* Respiratory Risk Assessment in Catalan Surgical Patients (ARISCAT) Criteria Low or Moderate Risk

Exclusion Criteria:

* Symptoms of upper respiratory tract infection or pulmonary infection in the past 4 weeks, chest X-ray suggests pneumonia
* Severe circulatory disease
* Children with bullae
* Intraoperative arterial blood pressure monitoring cannot be performed
* Respiratory Risk Assessment in Catalan Surgical Patients (ARISCAT) Criteria Rated High Risk

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complication(PPCs) rate at 7 days | 7 days after surgery
  PPCs are classified into 5 grades according to Postoperative pulmonary complications score fo JAMA.
  Grade 1:Cough, dry.Microatelectasis.Dyspnea, not due to other documented cause
  Grade 2:Cough, productive, not due to other documented cause.Bronchospasm.Hypoxemia (SpO2 ≤ 90%) at room air.Atelectasis.Hypercarbia (PaCO2 > 50 mmHg), requiring treatment
  Grade 3:Pleural effusion, resulting in thoracentesis.Pneumonia.Pneumothorax.Noninvasive ventilation, strictly applied to those with all of the following: a) oxygen saturation(SpO2)lower than 92% under supplemental oxygen; b) need of supplemental oxygen >5 L/min; and RR ≥ 30 bpm .Re-intubation postoperative or intubation, period of ventilator dependence (non-invasive or invasive ventilation) ≤ 48 hours
  Grade 4:Ventilatory failure: postoperative ventilator dependence exceeding 48 hours, or reintubation with subsequent period of ventilator dependence exceeding 48 hours
  Grade 5:Death before hospital discharge

SECONDARY OUTCOMES:
Oxygenation Index | 5 minutes after tracheal intubation (T1), 5 minutes after OLV (T2), 1 hour after OLV (T3-1), 2 hours after OLV (T3-2), 3 hours after OLV (T3-3), 4 hours after one-lung ventilation (T3-4), 5 minutes after the end of surgery (T4)
  Arterial partial pressure of oxygen divided by inspired oxygen concentration(PaO2/FiO2).
Driving pressure | 5 minutes after tracheal intubation (T1), 5 minutes after OLV (T2), 1 hour after OLV (T3-1), 2 hours after OLV (T3-2), 3 hours after OLV (T3-3), 4 hours after one-lung ventilation (T3-4), 5 minutes after the end of surgery (T4)
  Driving pressure = Pplateau -PEEP
Lung dynamic compliance | 5 minutes after tracheal intubation (T1), 5 minutes after OLV (T2), 1 hour after OLV (T3-1), 2 hours after OLV (T3-2), 3 hours after OLV (T3-3), 4 hours after one-lung ventilation (T3-4),5 minutes after the end of surgery (T4)
  LCdyn = TV/(Pplat-PEEP)
Modified lung ultrasound score | Postoperative 1 hour
  The score is calculated by adding up the 12 individual quadrant scores assessed using lung ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Children's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and with no end date
Access Criteria: Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal.
  Proposals should be directed to Dr Jiaxiang Chen; e mail address:cjxanes@163.com
  To gain access, data requestors will need to sign a data Access agreement.

REFERENCES:
- [Result] Costa Leme A, Hajjar LA, Volpe MS, Fukushima JT, De Santis Santiago RR, Osawa EA, Pinheiro de Almeida J, Gerent AM, Franco RA, Zanetti Feltrim MI, Nozawa E, de Moraes Coimbra VR, de Moraes Ianotti R, Hashizume CS, Kalil Filho R, Auler JO Jr, Jatene FB, Gomes Galas FR, Amato MB. Effect of Intensive vs Moderate Alveolar Recruitment Strategies Added to Lung-Protective Ventilation on Postoperative Pulmonary Complications: A Randomized Clinical Trial. JAMA. 2017 Apr 11;317(14):1422-1432. doi: 10.1001/jama.2017.2297. PMID 28322416
- [Result] Templeton TW, Miller SA, Lee LK, Kheterpal S, Mathis MR, Goenaga-Diaz EJ, Templeton LB, Saha AK; Multicenter Perioperative Outcomes Group Investigators. Hypoxemia in Young Children Undergoing One-lung Ventilation: A Retrospective Cohort Study. Anesthesiology. 2021 Nov 1;135(5):842-853. doi: 10.1097/ALN.0000000000003971. PMID 34543405
- [Result] Chandler D, Mosieri C, Kallurkar A, Pham AD, Okada LK, Kaye RJ, Cornett EM, Fox CJ, Urman RD, Kaye AD. Perioperative strategies for the reduction of postoperative pulmonary complications. Best Pract Res Clin Anaesthesiol. 2020 Jun;34(2):153-166. doi: 10.1016/j.bpa.2020.04.011. Epub 2020 Apr 23. PMID 32711826
- [Result] iPROVE Network investigators; Belda J, Ferrando C, Garutti I. The Effects of an Open-Lung Approach During One-Lung Ventilation on Postoperative Pulmonary Complications and Driving Pressure: A Descriptive, Multicenter National Study. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2665-2672. doi: 10.1053/j.jvca.2018.03.028. Epub 2018 Mar 27. PMID 29709437
- [Result] Lee JH, Ji SH, Lee HC, Jang YE, Kim EH, Kim HS, Kim JT. Evaluation of the intratidal compliance profile at different PEEP levels in children with healthy lungs: a prospective, crossover study. Br J Anaesth. 2020 Nov;125(5):818-825. doi: 10.1016/j.bja.2020.06.046. Epub 2020 Jul 15. PMID 32682552
- [Result] Xu D, Wei W, Chen L, Li S, Lian M. Effects of different positive end-expiratory pressure titrating strategies on oxygenation and respiratory mechanics during one- lung ventilation: a randomized controlled trial. Ann Palliat Med. 2021 Feb;10(2):1133-1144. doi: 10.21037/apm-19-441. Epub 2020 Sep 15. PMID 32954753
- [Result] Zhou ZF, Fang JB, Wang HF, He Y, Yu YJ, Xu Q, Ge YF, Zhang MZ, Hu SF. Effects of intraoperative PEEP on postoperative pulmonary complications in high-risk patients undergoing laparoscopic abdominal surgery: study protocol for a randomised controlled trial. BMJ Open. 2019 Oct 30;9(10):e028464. doi: 10.1136/bmjopen-2018-028464. PMID 31672709
- [Result] Lee JH, Bae JI, Jang YE, Kim EH, Kim HS, Kim JT. Lung protective ventilation during pulmonary resection in children: a prospective, single-centre, randomised controlled trial. Br J Anaesth. 2019 May;122(5):692-701. doi: 10.1016/j.bja.2019.02.013. Epub 2019 Mar 8. PMID 30916035
- [Result] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Result] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Result] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Result] Pereira SM, Tucci MR, Morais CCA, Simoes CM, Tonelotto BFF, Pompeo MS, Kay FU, Pelosi P, Vieira JE, Amato MBP. Individual Positive End-expiratory Pressure Settings Optimize Intraoperative Mechanical Ventilation and Reduce Postoperative Atelectasis. Anesthesiology. 2018 Dec;129(6):1070-1081. doi: 10.1097/ALN.0000000000002435. PMID 30260897
- [Derived] Chen J, Lin R, Shi X, Liang C, Hu W, Ma X, Xu L. Effects of individualised lung-protective ventilation with lung dynamic compliance-guided positive end-expiratory pressure titration on postoperative pulmonary complications of paediatric video-assisted thoracoscopic surgery: protocol for a randomised controlled trial. BMJ Paediatr Open. 2024 Jul 16;8(1):e002359. doi: 10.1136/bmjpo-2023-002359. PMID 39019541